CLINICAL TRIAL: NCT00440141
Title: Brimonidine 0.1% Versus Brinzolamide 1% as Adjunctive Therapy to Latanoprost 0.005%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MA-AP01
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2008-01-02 (Estimated); Status verified 2007-12

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost; Ophthalmic Solutions; Brimonidine Tartrate; brinzolamide

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: latanoprost 0.005% eye drops and brimonidine 0.1% eye drops
- 2 (Active Comparator)
  Interventions: Drug: latanoprost 0.005% eye drops and brinzolamide 1.0% eye drops

INTERVENTIONS:
Drug: latanoprost 0.005% eye drops and brimonidine 0.1% eye drops — latanoprost 0.005%, 1 drop nightly for 3 months and brimonidine 0.1% three-times daily for 3 months
  Other Names: Xalatan®; Alphagan® P
  Arms: 1
Drug: latanoprost 0.005% eye drops and brinzolamide 1.0% eye drops — latanoprost 0.005% 1 drop nightly for 3 months AND brinzolamide 1.0% 1% three-times daily for 3 months
  Other Names: Xalatan®; Azopt®
  Arms: 2

SUMMARY:
Patients with glaucoma or ocular hypertension currently being treated with latanoprost 0.005%, and in need of additional IOP lowering will be randomized to receive either brimonidine 0.1% or brinzolamide 1% three-times daily as adjunctive therapy to latanoprost 0.005%

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma or ocular hypertension in both eyes
* Currently being treated with latanoprost 0.005% QD
* IOP greater than or equal to 18mm Hg on latanoprost 0.005%
* Best-corrected VA of 20/200 or better in each eye
* Visual field within 6 months of study entry

Exclusion Criteria:

* Secondary glaucoma
* Active intraocular inflammation or macular edema
* Intraocular surgery or laser surgery within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
IOP | Month 3

SECONDARY OUTCOMES:
Tolerability | Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Director — Allergan
Locations (1):
- Atlanta, Georgia, United States

REFERENCES:
- [Derived] Day DG, Hollander DA. Brimonidine purite 0.1% versus brinzolamide 1% as adjunctive therapy to latanoprost in patients with glaucoma or ocular hypertension. Curr Med Res Opin. 2008 May;24(5):1435-42. doi: 10.1185/030079908x301848. Epub 2008 Apr 9. PMID 18402717